CLINICAL TRIAL: NCT04766710
Title: Implementation and Evaluation of a Community-Based Model for Delivery of Antiretroviral Therapy in Cambodia: A Quasi-Experimental Study
Brief Title: Community-Based Model for Delivery of Antiretroviral Therapy in Cambodia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: KHANA Center for Population Health Research (Other)
Responsible Party: Principal Investigator, Siyan Yi, Assistant Professor, National University of Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 030_PV_KHANA
Record Dates: First submitted 2021-01-15; First posted 2021-02-23 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections; AIDS
Keywords: HIV; Community-based services; ART; Operational research; Intervention; Cambodia
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This quasi-experimental study will consist of two arms. People living with HIV in the intervention arm will receive services from the CAD model, and those in the control arm will receive the standard prevention, care, and support services. The investigators will compare the outcome between these two arms.
Who Masked: Outcomes Assessor
Masking Description: Project coordinators and people living with HIV in the selected operational districts will not be masked to the intervention. However, all activities will be done without reference to the intervention group. The data analysts will be masked to intervention allocation and will only analyze de-identified data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based ART delivery (CAD) (Experimental): The CAD model intervention will take place for 24 months. A total of 2000 registered stable people living with HIV will form into the CAD group. The investigators have developed the implementation guide, monitoring tools, quality assurance checklist, and lists of people living with HIV in selected ART clinics for the CAD model intervention. The first step will be to extract the data disaggregated by gender, age, and type of sub-populations, including adolescents, female entertainment workers, men who have sex with men, transgender women, and people who use drugs from the national database using the definitions introduced by the WHO. Once the list is completed with patient ART codes, a consultative meeting combined with the project orientation will be convened. Providers from the selected ART clinics and implementing partners at each site will divide stable people living with HIV into their respective groups based on the ART sites.
  Interventions: Other: Community-based ART delivery (CAD)
- ART multi-month dispensing (MMD) (Active Comparator): A total of 2000 registered stable people living with HIV will form into the control group and received standard services under the MDD model. The control-arm participants will visit the ART clinics and collect their ARVs from the facility-based staff.
  Interventions: Other: ART multi-month dispensing (MMD)

INTERVENTIONS:
Other: Community-based ART delivery (CAD) — The frontline workers to implement the CAD model intervention will be people living with HIV recruited from the community who will plays roles as CAWs. The CAWs will receive intensive training, coaching, and mentoring from their respective ART clinics and implementing partners' field staff on ARV dispensing, drug storage, patient's vital sign assessment and recording, HIV education and counseling, medication adherence, referral systems, mental health, stigma and discrimination, and sexual and reproductive health of people living with HIV. To closely monitor the work of the CAWs, a respective ART clinic team, consisting of an ART counselor and a physician, will be tasked to conduct regular supervision along with the program team of the implementing partners to the community groups at least once a month in the first six months. After the six months, supervisory visits will be extended to once every two months.
  Arms: Community-based ART delivery (CAD)
Other: ART multi-month dispensing (MMD) — The control arm participants will receive routine services under the MMD model based on standard community-based prevention, care, and support practices in Cambodia. The NCHADS has introduced MDD in all ART sites across the country. However, so far, not all ART sites currently operate the MMD. The MMD is designed to help ART service providers implement MMD for eligible patients-that is, patients whose condition is determined to be stable-which will reduce the need for frequent visits and providers' workload. Stable people living with HIV receive care and support from counselors and ARVs at the clinics every four to six months.
  Arms: ART multi-month dispensing (MMD)

SUMMARY:
The community-based ART delivery (CAD) model will build on the existing framework to engage community action, operationalized in the current Global Fund-supported project. Community Action Workers (CAW), who are assigned to ART centers and conduct outreach work, are well-suited to administer CAD scheme. KHANA and the project partners all have implementation roles in the Global Fund-supported project and established working channels with the CAW.

While the previous experiences suggest the CAD model's effectiveness, implementing it in Cambodia requires adaptation to its specific local context. The proposed project will be implemented as an implementation study in nine ART sites and supported by a concrete evaluation plan. KHANA Center for Population Health Research will lead the research component.

The project has three strategic areas and corresponding deliverables as follows:

A. The development of a locally-fitted model: bringing ART closer to the people living with HIV B. The research: formulation, evaluation, documentation, and dissemination of the evidence, knowledge, and lessons learned C. The scale-up: advocacy for the SOP development to replicate/scale-up the CAD model

The project will benefit a wide range of stakeholders. The approximately 2,000 ART clients enrolled in the nine selected clinics will face less cost, time, and discrimination, which will also benefit their families. The clinics will have a reduced workload on site, and they would be able to improve the quality of care for the visiting clients. The Cambodian health system will obtain a CAD model tailored to the country's local context and develop Standard Operating Procedures for the scheme with readily involved stakeholders. The scale-up of the model will benefit all other ART clinics and clients in the country.

The 36-months project starting from June 1, 2019, will include six months of start-up and baseline assessments, 24-month intervention, and six-month evaluation.

DETAILED DESCRIPTION:
One of the challenges in the Cambodian HIV response is the relatively low rate of retention in care and viral load suppression among people living with HIV on ART. According to a report from the National Center for HIV/AIDS, Dermatology and STD (NCHADS), by the end of September 2017, approximately 98% (n= 58,268) of people living with HIV diagnosed in the whole country were initiated on ART. Of them, 75% were virally suppressed, and 89% were retained on the treatment 12 months after the treatment initiation. Similarly, a recent study conducted by KHANA Center for Population Research in 11 ART clinics across the country found that the rate of viral suppression among adolescents living with HIV aged 15-17 was 76.8%.

To date, ART in Cambodia has been administered only at the government ART clinics. Nationally, there are 66 ART Clinics in 22 of the 25 provinces. Making a trip to an ART clinic on a monthly or bimonthly basis to receive repeated prescriptions poses a heavy burden on the clients in terms of both time and money. Besides, as the Global Fund Funding Request points out (pp.7-8), besides self-stigma, people living with HIV and key populations continue to face stigma and discrimination in their communities, in accessing health and other services, and at the household level. Furthermore, under the current scheme, the necessity for the ART clinics to meet the demand of all of the ART clients, including the stable clients who visit bi-monthly, is a huge burden on the facilities and the service providers. Fewer client visits per given timeframe are expected to help the health workers spend more time per visiting client and improve the service quality.

Community-based service delivery has been an integral part of the response to HIV in other parts of the world. Cambodia's national HIV program acknowledges the major contribution of such an approach, including the proposed CAD model. In 2016, the World Health Organization (WHO) recommended that stable ART clients can safely reduce the frequency of clinic visits, potentially receiving ART in community settings. Researches from other contexts have also suggested that communities can be engaged to provide ART with good outcomes. Most CAD models have been demonstrated to reduce burdens for patients and the health systems, increased retention in care, and lower service provider costs. KHANA and its partners, including NCHADS, believe that an adaptation of an ART delivery model that meaningfully includes community-based services will be essential, particularly as the national program intensifies case-finding and the "Treat All" approach, to meet the national targets.

KHANA has been a leader of the country's community-led HIV response and was one of the key members in developing the "Consolidated Operational Framework on Community Action Approach to Implement B-IACM towards achieving 90-90-90 in Cambodia (Community Action Framework)" of NCHADS. For the past 20 years, KHANA has supported the capacity building of the HIV-affected communities, who now bring invaluable contributions to the design of the HIV response in Cambodia. The Community Action Framework aims to ensure the continued participation of the communities, thus strengthening the health system and empowering the HIV-affected communities. The current Global Fund-supported project applies this framework to detect undiagnosed people living with HIV by promoting HIV testing and counseling in the communities and improve the HIV care cascade. KHANA sees an opportunity to extend this framework's application in the form of CAD with the support of the 5% Initiative.

The Community Action Framework has a section on CAD; however, there is a need to operationalize this model and demonstrating its applicability in the Cambodian context. The proposed project will develop a CAD model considering the evidence and findings of previous studies, the Cambodian local context, and the principles set by the national HIV program. As an operational research project, it will be implemented to reach approximately 2,000 people living with HIV who are categorized as 'stable' (on ART for 12 months or more, clinically stable, undetectable viral load) in nine selected ART clinics, five urban and four rural, in the five provinces. In total, 82 community-based ART groups will be established, with approximately 25 members in each group. The designated CAW will coordinate the groups with technical support from five project assistants, one per province.

In the architecture of the current Global Fund-supported project, the Community-Based Prevention, Care and Support (CBPCS) are implemented for people living with HIV in greatest needs and other target populations by civil society organization (CSO) workers at the ART clinics; i.e., Community Action Counsellors (CAC), Facility-Based Workers (FBW) and CAW. They will contribute to the daily facility activities and perform outreach work as needed. CAWs are assigned to 37 ART sites, and their responsibilities will include: a) provision of case management and support for people living with HIV in greatest needs (e.g., people living with HIV who are newly enrolled in ART, pregnant women, children under five years and adolescents) to improve drug adherence, missed appointment issues or treatment failure and b) being in contact with Village Health Support Groups (VHSG) to encourage HIV testing and counseling and trace new cases. The administration of CAD fits well in the function of CAW.

The project is strategized around three key areas as follows:

1. Bringing ART closer to the people living with HIV This innovative CAD model's main concept is that the community-based ART provision brings the treatment to come closer to people living with HIV. It is made possible by CAW who bring pre-packed ARV refill and various support services to the members of Community ART Groups. A technology-based tool using tablets will be introduced to the CAW as educational materials and monitoring tools.

   Accessibility of ARV distribution points is crucial to the success of this scheme. Therefore, the distribution points will be located at the monthly meeting sites of the local self-help groups. Stable ART clients who are members of the scheme will visit the designated ART clinic for consultation and viral load monitoring every six months. The project will also work to reactivate the existing savings initiative within such self-help groups to contribute to such community groups' sustainability.

   Linkages with the designated ART clinics will be strengthened through capacity-building activities, coaching, and mentoring. Training will be provided to the relevant ART clinic staff members on the new CAD model's overall objectives and on the roles they will play in the project implementation.

   Gender, age, and populations are parameters that are expected to determine the effectiveness of the model significantly. The project will have mixed-gender groups and population-specific groups (e.g., male, female, transgender women, men who have sex with men). The project design will also consider the special needs of different population groups such as female entertainment workers (FEWs) and lesbian, gay, bisexual, transgender, and intersex (LGBTI) more broadly.
2. Evaluation, documentation, and dissemination of the project findings and lessons learned

The project will provide an opportunity to generate various program findings, evidence and lessons learned, which will be documented and disseminated through:

* Routine data collection for project monitoring and harmonization with/integration into the B-IACM approach and national ART database system.
* Case study documentation per site and comparative analyses.
* Presentations at national HIV/AIDS Technical Working Group meetings to support knowledge sharing and replication of the model.
* Dissemination of the findings nationally to the Ministry of Health and other national and international stakeholders to inform evidence-based policy dialogues.
* Presentations at national, regional, and international scientific conferences.
* Operational reports and international peer-reviewed publications.

ELIGIBILITY:
Inclusion criteria:

1. Receiving ART for at least one year.
2. No adverse drug reactions or ARV drug interactions requiring regular monitoring.
3. No suspected or confirmed tuberculosis, no other opportunistic infections, and not on any prophylaxis.
4. Not pregnant/breastfeeding (for women).
5. Having a good understanding of lifelong treatment and adherence to the medication.
6. Presenting with evidence of treatment success: two consecutive undetectable viral load measures (or, in the absence of viral load monitoring, CD4 counts above 200 cells/mm3 and objective adherence measure).
7. Aged ≥15 years.
8. On the first-line ARV regimen.

Exclusion criteria

1. Unstable people living with HIV as defined above
2. Mobile populations

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4102 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Percent of people living with HIV with viral suppression | 24 months after the intervention started
  Viral load At least 90% of participants in intervention arm will have a viral load <1000 RNA copies/mL by the endline of the intervention
Percent of people living with HIV who remained in HIV care and treatment | 24 months after the intervention started
  At least 90% of participants in the intervention will be retained in care and treatment 12 months after the treatment started
Percent of people living with HIV with good adherence to ART | 24 months after the intervention started
  At least 90% of the participants in the intervention will report good adherence to ART at the endline.
Percent of healthcare providers at ART clinics who reported reduced workload | 24 months after the intervention started
  Workload at ART clinics will be self-reported by health care workers providing ART services at the clinics. The investigators hypothesize that a significantly higher proportion of health care providers at ART clinics under the CAD intervention arm will agree that their workload has been reduced at endline compared to baseline.

SECONDARY OUTCOMES:
Cost-effectiveness of community-based ART delivery (CAD) model intervention | 24 months after the intervention started
  For the cost-effectiveness analyses, direct and indirect medical costs for follow-up care and ARV refills will be collected. The costs in this community-based ART delivery intervention will be compared with the costs in standard care services (facility-based and multi-month dispensing model). The investigators anticipated that the community-based ART delivery intervention will be similar in all intervention and service delivery models. However, CAD model will help save time and costs of people living with HIV in the intervention arm.
Percent of people living with HIV who reported improved quality of life | 24 months after the intervention started
  The quality of life of people living with HIV will be measured using WHO's Quality of Life HIV brief questionnaire (WHOQOL-HIV-BREF). The scale's domain score ranges from 4 to 20. Higher scores indicate a better quality of life. The investigators hypothesized that the proportion of people living with HIV who reported a higher quality of life would increase more significantly from baseline to endline among participants in the community-based ART delivery (CAD) intervention arm than those in the control arm.
Percent of people living with HIV who reported improved mental health | 24 months after the intervention started
  The mental health of people living with HIV will be measured using the Center for Epidemiologic Studies Depression Scale (CES-D). The total CES-D score ranges from 0 to 60. A subject with a CES-D score of ≥16 will be defined as having depressive symptoms. The investigators hypothesized that the proportion of people living with HIV who reported having depressive symptoms would decrease more significantly from baseline to endline among participants in the community-based ART delivery (CAD) intervention arm than in the control arm.
Percent of people living with HIV who reported improved social support health | 24 months after the intervention started
  Social support for people living with HIV will be measured using Berlin Social Support Scale (BSSS). The BSSS's total score ranges from 15 to 60, with higher scores indicating higher social support. The investigators hypothesized that the proportion of people living with HIV who perceived a high social support level would increase more significantly from baseline to endline among participants in the community-based ART delivery (CAD) intervention arm than those in the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sok Chamreun Choub, MA, Study Chair — KHANA Center for Population Health Research; Penh Sun Ly, MD, Study Chair — National Center for HIV, Dermatology and STD
Locations (3):
- Cambodia (3):
  - KHANA Center for Population Health Research, Phnom Penh
  - Cambodia Anti-Tuberculosis Association, Phnom Penh
  - National Center for Tuberculosis and Leprosy Control, Phnom Penh

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study will be available from the principal investigator on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will permanently available after the main report of the project has been published.

REFERENCES:
- [Background] Tuot S, Teo AKJ, Cazabon D, Sok S, Ung M, Ly S, Choub SC, Yi S. Acceptability of active case finding with a seed-and-recruit model to improve tuberculosis case detection and linkage to treatment in Cambodia: A qualitative study. PLoS One. 2019 Jul 2;14(7):e0210919. doi: 10.1371/journal.pone.0210919. eCollection 2019. PMID 31265458
- [Result] Chhim K, Mburu G, Tuot S, Sopha R, Khol V, Chhoun P, Yi S. Factors associated with viral non-suppression among adolescents living with HIV in Cambodia: a cross-sectional study. AIDS Res Ther. 2018 Nov 17;15(1):20. doi: 10.1186/s12981-018-0205-z. PMID 30445984
- [Result] Rivers PA, Glover SH. Health care competition, strategic mission, and patient satisfaction: research model and propositions. J Health Organ Manag. 2008;22(6):627-41. doi: 10.1108/14777260810916597. PMID 19579575
- [Result] Moudachirou R, Van Cutsem G, Chuy RI, Tweya H, Senkoro M, Mabhala M, Zolfo M. Retention and sustained viral suppression in HIV patients transferred to community refill centres in Kinshasa, DRC. Public Health Action. 2020 Mar 21;10(1):33-37. doi: 10.5588/pha.19.0067. PMID 32368522
- [Result] Mutasa-Apollo T, Ford N, Wiens M, Socias ME, Negussie E, Wu P, Popoff E, Park J, Mills EJ, Kanters S. Effect of frequency of clinic visits and medication pick-up on antiretroviral treatment outcomes: a systematic literature review and meta-analysis. J Int AIDS Soc. 2017 Jul 21;20(Suppl 4):21647. doi: 10.7448/IAS.20.5.21647. PMID 28770599
- [Result] Chaiyachati KH, Ogbuoji O, Price M, Suthar AB, Negussie EK, Barnighausen T. Interventions to improve adherence to antiretroviral therapy: a rapid systematic review. AIDS. 2014 Mar;28 Suppl 2:S187-204. doi: 10.1097/QAD.0000000000000252. PMID 24849479
- [Result] Yi S, Chhoun P, Suong S, Thin K, Brody C, Tuot S. AIDS-related stigma and mental disorders among people living with HIV: a cross-sectional study in Cambodia. PLoS One. 2015 Mar 25;10(3):e0121461. doi: 10.1371/journal.pone.0121461. eCollection 2015. PMID 25806534
- [Result] Bemelmans M, Baert S, Goemaere E, Wilkinson L, Vandendyck M, van Cutsem G, Silva C, Perry S, Szumilin E, Gerstenhaber R, Kalenga L, Biot M, Ford N. Community-supported models of care for people on HIV treatment in sub-Saharan Africa. Trop Med Int Health. 2014 Aug;19(8):968-77. doi: 10.1111/tmi.12332. Epub 2014 May 28. PMID 24889337
- [Result] Okoboi S, Ding E, Persuad S, Wangisi J, Birungi J, Shurgold S, Kato D, Nyonyintono M, Egessa A, Bakanda C, Munderi P, Kaleebu P, Moore DM. Community-based ART distribution system can effectively facilitate long-term program retention and low-rates of death and virologic failure in rural Uganda. AIDS Res Ther. 2015 Nov 12;12:37. doi: 10.1186/s12981-015-0077-4. eCollection 2015. PMID 26566390
- [Result] Decroo T, Koole O, Remartinez D, dos Santos N, Dezembro S, Jofrisse M, Rasschaert F, Biot M, Laga M. Four-year retention and risk factors for attrition among members of community ART groups in Tete, Mozambique. Trop Med Int Health. 2014 May;19(5):514-21. doi: 10.1111/tmi.12278. Epub 2014 Feb 12. PMID 24898272
- [Result] Faturiyele IO, Appolinare T, Ngorima-Mabhena N, Fatti G, Tshabalala I, Tukei VJ, Pisa PT. Outcomes of community-based differentiated models of multi-month dispensing of antiretroviral medication among stable HIV-infected patients in Lesotho: a cluster randomised non-inferiority trial protocol. BMC Public Health. 2018 Aug 29;18(1):1069. doi: 10.1186/s12889-018-5961-0. PMID 30157896
- [Result] Decroo T, Telfer B, Dores CD, White RA, Santos ND, Mkwamba A, Dezembro S, Joffrisse M, Ellman T, Metcalf C. Effect of Community ART Groups on retention-in-care among patients on ART in Tete Province, Mozambique: a cohort study. BMJ Open. 2017 Aug 11;7(8):e016800. doi: 10.1136/bmjopen-2017-016800. PMID 28801427
- [Result] Decroo T, Rasschaert F, Telfer B, Remartinez D, Laga M, Ford N. Community-based antiretroviral therapy programs can overcome barriers to retention of patients and decongest health services in sub-Saharan Africa: a systematic review. Int Health. 2013 Sep;5(3):169-79. doi: 10.1093/inthealth/iht016. Epub 2013 Jul 30. PMID 24030268
- [Result] Rand CS. Measuring adherence with therapy for chronic diseases: implications for the treatment of heterozygous familial hypercholesterolemia. Am J Cardiol. 1993 Sep 30;72(10):68D-74D. doi: 10.1016/0002-9149(93)90014-4. PMID 8213501
- [Result] Jay S, Litt IF, Durant RH. Compliance with therapeutic regimens. J Adolesc Health Care. 1984 Apr;5(2):124-36. doi: 10.1016/s0197-0070(84)80012-1. PMID 6368505
- [Result] Murray KR, Dulli LS, Ridgeway K, Dal Santo L, Darrow de Mora D, Olsen P, Silverstein H, McCarraher DR. Improving retention in HIV care among adolescents and adults in low- and middle-income countries: A systematic review of the literature. PLoS One. 2017 Sep 29;12(9):e0184879. doi: 10.1371/journal.pone.0184879. eCollection 2017. PMID 28961253
- [Result] Rasschaert F, Decroo T, Remartinez D, Telfer B, Lessitala F, Biot M, Candrinho B, Van Damme W. Adapting a community-based ART delivery model to the patients' needs: a mixed methods research in Tete, Mozambique. BMC Public Health. 2014 Apr 15;14:364. doi: 10.1186/1471-2458-14-364. PMID 24735550
- [Result] Ibrahim AA, Akindele MO, Ganiyu SO, Kaka B, Abdullahi BB, Sulaiman SK, Fatoye F. The Hausa 12-item short-form health survey (SF-12): Translation, cross-cultural adaptation and validation in mixed urban and rural Nigerian populations with chronic low back pain. PLoS One. 2020 May 7;15(5):e0232223. doi: 10.1371/journal.pone.0232223. eCollection 2020. PMID 32379769
- [Derived] Yam LYE, Chhoun P, Tian Z, Nagashima-Hayashi M, Zahari M, Tuot S, Samreth S, Ngauv B, Ouk V, Prem K, Yi S. Cost-effectiveness analysis of a community-based model for delivery of antiretroviral therapy to people with clinically stable HIV in Cambodia. J Int AIDS Soc. 2025 Jul;28 Suppl 3(Suppl 3):e26476. doi: 10.1002/jia2.26476. PMID 40623943
- [Derived] Tuot S, Teo AKJ, Prem K, Chhoun P, Pall C, Ung M, Ly PS, Jimba M, Yi S. Community-based model for the delivery of antiretroviral therapy in Cambodia: a quasi-experimental study protocol. BMC Infect Dis. 2021 Aug 6;21(1):763. doi: 10.1186/s12879-021-06414-y. PMID 34362310